CLINICAL TRIAL: NCT00642902
Title: A Four-Arm Randomized, Double-Blind, Placebo-Controlled, Multicenter Phase II Study to Evaluate the Safety, Tolerability and Efficacy as Assessed by Frequent MRI Measures of 3 Doses of Atacicept Monotherapy in Subjects With Relapsing Multiple Sclerosis (RMS) Over a 36 Week Treatment Course
Brief Title: A Phase 2 Study of Atacicept in Subjects With Relapsing Multiple Sclerosis (ATAMS)
Acronym: ATAMS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor voluntarily decided to terminate trial due to increased MS disease activity in atacicept arms as compared to placebo during a routine IDMC review.
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 28063
Record Dates: First submitted 2008-03-21; First posted 2008-03-25 (Estimated); Results first posted 2016-05-24 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-04

CONDITIONS: Relapsing Multiple Sclerosis
Keywords: Relapsing Multiple Sclerosis; Atacicept
MeSH Terms: interventions — TACI receptor-IgG Fc fragment fusion protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Atacicept 25 mg (Experimental)
  Interventions: Drug: Atacicept
- Atacicept 75 mg (Experimental)
  Interventions: Drug: Atacicept
- Atacicept 150 mg (Experimental)
  Interventions: Drug: Atacicept
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo matched to atacicept

INTERVENTIONS:
Drug: Atacicept — Atacicept will be administered subcutaneously at a dose of 25 milligram (mg) twice a week for initial 4 weeks as loading dose, followed by 25 mg once a week for subsequent 32 weeks.
  Arms: Atacicept 25 mg
Drug: Atacicept — Atacicept will be administered subcutaneously at a dose of 75 mg twice a week for initial 4 weeks as loading dose, followed by 75 mg once a week for subsequent 32 weeks.
  Arms: Atacicept 75 mg
Drug: Atacicept — Atacicept will be administered subcutaneously at a dose of 150 mg twice a week for initial 4 weeks as loading dose, followed by 150 mg once a week for subsequent 32 weeks.
  Arms: Atacicept 150 mg
Drug: Placebo matched to atacicept — Placebo matched to atacicept will be administered subcutaneously twice a week for initial 4 weeks, followed by once a week for subsequent 32 weeks.
  Arms: Placebo

SUMMARY:
To evaluate the safety and tolerability of atacicept and to explore if atacicept reduces central nervous system inflammation in subjects with relapsing multiple sclerosis (RMS) as assessed by frequent magnetic resonance imaging (MRI). This study is randomised. Study medication is administered via subcutaneous (under the skin) injections.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosis of RMS (as per McDonald criteria, 2005) Other protocol-defined inclusion criteria could apply.

Exclusion Criteria:

* Have primary progressive multiple sclerosis (MS)
* Have secondary progressive MS without superimposed relapses
* Relevant cardiac, hepatic and renal diseases as specified in the protocol
* Pretreatment with immunosuppressants and immunomodulating drugs as specified in the protocol
* Clinical significant abnormalities in blood cell counts and immunoglobulin levels as specified in the protocol
* Clinical significant acute or chronic infections as specified in the protocol Other protocol-defined exclusion criteria could apply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 255 (Actual)
Dates: Start 2008-04; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono, an affiliate of Merck KGaA Darmstadt, Germany
Locations (50):
- United States (8):
  - Research Site, Phoenix, Arizona
  - Research Site, Atlanta, Georgia
  - Research Site, Northbrook, Illinois
  - Research Site, East Lansing, Michigan
  - Research Site, Jefferson, New Hampshire
  - Research Site, Cleveland, Ohio
  - Philadelphia, Pennsylvania
  - Research Site, Nashville, Tennessee
- Australia (4):
  - Research Site, Box Hill
  - Research Site, Fitzroy
  - Research Site, New Lambton
  - Research Site, Woodville
- Research Site, Innsbruck, Austria
- Belgium (2):
  - Research Site, Diepenbeek
  - Research Site, Sijsele
- Canada (3):
  - Research Site, Calgary, Alberta
  - Research Site, Ottawa, Ontario
  - Research Site, Ontario
- Czechia (3):
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Olomouc
- France (2):
  - Research Site, Caen
  - Research Site, Saint-Herblain
- Germany (2):
  - Research Site, Bochum
  - Research Site, Düsseldorf
- Research Site, Beirut, Lebanon
- Research Site, Kaunas, Lithuania
- Netherlands (3):
  - Research Site, Breda
  - Research Site, Nieuwegein
  - Research Site, Rotterdam
- Russia (8):
  - Research Site, Dnipropetrovsk
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Saint Petersburg
  - Research Site, Samara
  - Research Site, Vladimir
  - Research Site, Yaroslavl
  - Research Site, Yekaterinburg
- Spain (3):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Málaga
- Research Site, Stockholm, Sweden
- Research Site, Basel, Switzerland
- Ukraine (4):
  - Research Site, Kharkiv
  - Research Site, Kyiv
  - Research Site, Odesa
  - Research Site, Uzhhorod
- United Kingdom (3):
  - Research Site, London
  - Research Site, Sheffield
  - Research Site, Stoke-on-Trent

REFERENCES:
- [Derived] Kappos L, Hartung HP, Freedman MS, Boyko A, Radu EW, Mikol DD, Lamarine M, Hyvert Y, Freudensprung U, Plitz T, van Beek J; ATAMS Study Group. Atacicept in multiple sclerosis (ATAMS): a randomised, placebo-controlled, double-blind, phase 2 trial. Lancet Neurol. 2014 Apr;13(4):353-63. doi: 10.1016/S1474-4422(14)70028-6. Epub 2014 Mar 6. PMID 24613349
- See also: Related Info — http://www.mslifelines.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo matched to atacicept was administered subcutaneously twice a week for initial 4 weeks, followed by once a week for subsequent 32 weeks.
- Atacicept 25 mg: Atacicept was administered subcutaneously at a dose of 25 milligram (mg) twice a week for initial 4 weeks as loading dose, followed by 25 mg once a week for subsequent 32 weeks.
- Atacicept 75 mg: Atacicept was administered subcutaneously at a dose of 75 mg twice a week for initial 4 weeks as loading dose, followed by 75 mg once a week for subsequent 32 weeks.
- Atacicept 150 mg: Atacicept was administered subcutaneously at a dose of 150 mg twice a week for initial 4 weeks as loading dose, followed by 150 mg once a week for subsequent 32 weeks.
Period: Overall Study
Arm/Group | Placebo | Atacicept 25 mg | Atacicept 75 mg | Atacicept 150 mg
Started | 63 | 63 | 64 | 65
Treated | 63 | 63 | 63 | 65
Completed | 23 | 21 | 21 | 25
Not Completed | 40 | 42 | 43 | 40
Not completed — Adverse Event | 0 | 1 | 3 | 1
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 3 | 3 | 0
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Premature termination of clinical trial | 37 | 32 | 35 | 35
Not completed — Randomized, but not treated | 0 | 0 | 1 | 0
Not completed — Other | 1 | 5 | 1 | 4

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Atacicept 25 mg | Atacicept 75 mg | Atacicept 150 mg | Total
Number analyzed (Participants) | 63 | 63 | 64 | 65 | 255
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (10.5) | 37.5 (8.5) | 38.0 (10.1) | 37.5 (10.5) | 37.7 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 34 | 44 | 46 | 169
  Male | 18 | 29 | 20 | 19 | 86

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Time Constant 1 (T1) Gadolinium (Gd)-Enhancing Lesions Per Participant Per Scan
Description: Analysis of T1 Gd-enhancing lesions was done using magnetic resonance imaging (MRI) scans. Only post-baseline scans were included in the calculation of this endpoint (excluding the Study Day 1 scan which had been conducted before first dosing).
Time Frame: Weeks 12 to 36
Population: ITT population included all randomized participants.
Measure: Mean (95% Confidence Interval); unit: lesions/participant/scan
Arm/Group | Placebo | Atacicept 25 mg | Atacicept 75 mg | Atacicept 150 mg
Number analyzed (Participants) | 63 | 63 | 64 | 65
lesions/participant/scan | 3.07 [1.40 to 6.77] | 2.26 [0.97 to 5.27] | 2.30 [1.08 to 4.92] | 2.49 [1.18 to 5.27]

2. Secondary Outcome: Number of New T1 Gd-enhancing Lesions Per Participant
Description: Analysis of new T1 Gd-enhancing lesions was done using MRI scans.
Time Frame: Weeks 12, 24, 36
Population: ITT population included all randomized participants. 'n' signifies participants who were evaluable for this measure at given time points for each group, respectively.
Measure: Mean (Standard Deviation); unit: lesions/participant
Arm/Group | Placebo | Atacicept 25 mg | Atacicept 75 mg | Atacicept 150 mg
Number analyzed (Participants) | 63 | 63 | 64 | 65
lesions/participant
  Week 12 (n=55, 45, 50, 55) | 2.55 (7.95) | 2.71 (7.67) | 3.20 (6.41) | 2.96 (6.58)
  Week 24 (n=41, 34, 37, 41) | 0.83 (1.70) | 1.50 (2.79) | 1.54 (2.96) | 1.54 (2.94)
  Week 36 (n=23, 22, 24, 26) | 0.43 (0.90) | 1.68 (5.09) | 1.38 (1.93) | 0.54 (1.07)

3. Secondary Outcome: Percentage of Participants Free From Relapses
Description: A relapse was defined as the fulfillment of all the following criteria: a) neurological abnormality, either newly appearing or re-appearing, with abnormality specified by both i) neurological abnormality separated by at least 30 days from onset of a preceding clinical event, and ii) neurological abnormality lasting for at least 24 hours; b) absence of fever or known infection (fever with temperature [axillary, orally, or intrauriculary] greater than (>) 37.5 degrees Celsius or 99.5 degrees Fahrenheit); and c) objective neurological impairment, correlating with the participant's reported symptoms, defined as either i) increase in at least 1 of the functional systems of the Expanded Disability Status Scale (EDSS), or ii) increase of the total EDSS score. Percentage of participants free from relapses during 36-week treatment period was reported.
Time Frame: Baseline up to Week 36
Population: ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Atacicept 25 mg | Atacicept 75 mg | Atacicept 150 mg
Number analyzed (Participants) | 63 | 63 | 64 | 65
percentage of participants | 81.0 | 69.8 | 71.9 | 61.5

4. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An AE was defined as any new untoward medical occurrences/worsening of pre-existing medical condition without regard to possibility of causal relationship. An SAE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect. Treatment-emergent are events between first dose of study drug up to 12 weeks after the last dose of the study drug that were absent before treatment or that worsened relative to pretreatment state. Number of subjects with TEAEs included subjects with both non serious and serious TEAEs.
Time Frame: From the first dose of study drug administration up to 12 weeks after the last dose of the study drug
Population: Safety population included all participants who received at least 1 dose of treatment (either active or placebo).
Measure: Number; unit: participants
Arm/Group | Placebo | Atacicept 25 mg | Atacicept 75 mg | Atacicept 150 mg
Number analyzed (Participants) | 63 | 63 | 63 | 65
participants
  TEAEs | 46 | 40 | 39 | 52
  Serious TEAEs | 1 | 3 | 3 | 1

ADVERSE EVENTS:
Time Frame: From the first dose of study drug administration up to 12 weeks after the last dose of the study drug
Arm/Group | Placebo | Atacicept 25 mg | Atacicept 75 mg | Atacicept 150 mg
Serious Adverse Events (participants affected / at risk) | 1/63 | 3/63 | 3/63 | 1/65
Other Adverse Events (participants affected / at risk) | 33/63 | 30/63 | 34/63 | 44/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=63) | Atacicept 25 mg (N=63) | Atacicept 75 mg (N=63) | Atacicept 150 mg (N=65)
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Acute psychosis (Psychiatric disorders) | 0 | 1 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Lung abscess (Infections and infestations) | 0 | 0 | 1 | 0
Pyothorax (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 0
Body temperature decreased (Investigations) | 0 | 0 | 1 | 0
Otitis media acute (Infections and infestations) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=63) | Atacicept 25 mg (N=63) | Atacicept 75 mg (N=63) | Atacicept 150 mg (N=65)
Injection site reaction (General disorders) | 8 | 19 | 24 | 32
Fatigue (General disorders) | 0 | 1 | 3 | 4
Injection site pain (General disorders) | 2 | 2 | 0 | 4
Nasopharyngitis (Infections and infestations) | 6 | 4 | 7 | 13
Urinary tract infection (Infections and infestations) | 3 | 4 | 7 | 3
Upper respiratory tract infection (Infections and infestations) | 3 | 1 | 4 | 8
Bronchitis (Infections and infestations) | 1 | 2 | 1 | 5
Influenza (Infections and infestations) | 5 | 1 | 1 | 2
Headache (Nervous system disorders) | 11 | 8 | 3 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 3 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 3 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 3 | 5
Nausea (Gastrointestinal disorders) | 2 | 3 | 1 | 4

LIMITATIONS AND CAVEATS:
Sponsor voluntarily decided to prematurely terminate this trial due to an increase in multiple sclerosis (MS) disease activity observed in atacicept arms as compared to placebo during a routine independent data monitoring committee (IDMC) review.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to publishing results, Institution and Principal Investigator (PI) must first provide Sponsor with a copy of proposed publication for review at least 30 days prior to submission. If Institution and PI do not agree to modification, they shall so notify Sponsor and postpone submission for additional 60 days to allow Sponsor to seek legal remedies or file patent applications. There is a need for coordinated approach to any publication of results from sites for any multi-site study.